CLINICAL TRIAL: NCT06499142
Title: STP.168 Clinical Study Protocol Parakeet
Acronym: Parakeet
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovision Medical Products Inc (Industry)
Responsible Party: Principal Investigator, Christine Vergely, Director of Regulatory Affairs, Neurovision Medical Products Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STP.168
Record Dates: First submitted 2024-06-19; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Parathyroid; Anomaly; Parathyroid Dysfunction; Hyperparathyroidism; Parathyroid Gland Adenoma
Keywords: Immunoassay Lateral Flow, Parathyroid gland, PTH, FNA; Parathyroid gland,; PTH,; FNA
MeSH Terms: conditions — Congenital Abnormalities; Parathyroid Diseases; Hyperparathyroidism; Parathyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Parathyroidectomy (Experimental): Patients undergoing parathyroidectomy for Hyperparathyroidism
  Interventions: Device: Parakeet:The Parakeet Rapid Parathyroid Testing Kit is a rapid immunoassay designed to detect Parathormone (PTH) in a test sample.

INTERVENTIONS:
Device: Parakeet:The Parakeet Rapid Parathyroid Testing Kit is a rapid immunoassay designed to detect Parathormone (PTH) in a test sample. — The Parakeet Rapid Parathyroid Testing Kit is a rapid immunoassay designed to detect Parathormone (PTH) in a test sample. The Parakeet is a point of care test completely controlled by the surgeon and operating team. It uses the scientific principle of "Lateral Flow" of antibody-antigen-conjugate complexes being arrested in a "Test Line".

SUMMARY:
STUDY PURPOSE

The purpose of this study is to demonstrate the performance of the Parakeet Rapid Parathyroid Testing Kit by comparing Parakeet results with histopathologic Diagnosis.

STUDY OBJECTIVES

To demonstrate the positive percent agreement (PPA) and negative percent agreement (NPA) of the Parakeet Rapid Parathyroid Testing kit test results in FNA from excised tissue during parathyroid surgery with Pathologic Diagnosis.

DETAILED DESCRIPTION:
The Parakeet is a lateral flow cassette designed to aid in the detection of parathyroid gland by identifying tissue with parathyroid hormone levels > 60 pg./ml in a fine needle aspirate specimen. The FNA specimen of the target tissue is combined with running fluid and deposited into the sample well of a lateral flow cassette. Lateral flow occurs and the Test Line begins to darken within minutes if PTH is present in quantities > 60 pg./ml. At 5 minutes, a full visualization of the TL is done. A negative test (< 60 pg./ml of PTH in the sample) shows darkening of the Control Line only. Absence of Control Line development indicates a defective test kit.

INTENDED USE

The Parakeet Rapid Parathyroid Testing Kit is an immunoassay lateral flow cassette intended to detect qualitative differences in extracellular concentration of parathyroid hormone in excised samples suspected of being parathyroid glands as an adjunct to current clinical methods, including histopathology, to locate the parathyroid glands.

INDICATIONS FOR USE

The Parakeet Rapid Parathyroid Testing Kit is indicated for use in adult patients where location of the parathyroid glands is medically necessary, such as in patients undergoing parathyroidectomy for Hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

Men and women

≥18 years of age Scheduled for Parathyroid surgery

Exclusion Criteria:

Unable or unwilling to provide informed consent Subject has any condition that in the opinion of the investigator should preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The participant's IVD PTH concentration is < 57 pg/ml and the pathology report will be negative for parathyroid gland. The participant's IVD PTH concentration is > 57 pg/ml and the pathology report will be positive for parathyroid gland. | 5 minutes
  PT ID (visual): Visual Reading for FNA only; Positive (indicates a PTG), Negative (non-PTG). Qualitative variable, if the sample demonstrates a Test Line visual development, it is "Positive." If the Test Line does not demonstrate visual development this indicates less than the threshold of 60 pg./ml of PTH and it is considered negative (non-PTG) (Figure 5). The visual reading is by the tester and the surgeon is not notified. A faint or equivocal Test Line reading should be evaluated by the tester and repeated or other measures taken

CONTACTS AND LOCATIONS:
Overall Officials: Lee J Rea, Dr, Study Director — Neurovision Medical Product, Inc
Locations (1):
- Ventura County Medical center Santa Paula, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barczynski M, Branstrom R, Dionigi G, Mihai R. Sporadic multiple parathyroid gland disease--a consensus report of the European Society of Endocrine Surgeons (ESES). Langenbecks Arch Surg. 2015 Dec;400(8):887-905. doi: 10.1007/s00423-015-1348-1. Epub 2015 Nov 5. PMID 26542689
- [Background] Obolonczyk L, Karwacka I, Wisniewski P, Sworczak K, Oseka T. The Current Role of Parathyroid Fine-Needle Biopsy (P-FNAB) with iPTH-Washout Concentration (iPTH-WC) in Primary Hyperparathyroidism: A Single Center Experience and Literature Review. Biomedicines. 2022 Jan 6;10(1):123. doi: 10.3390/biomedicines10010123. PMID 35052802